CLINICAL TRIAL: NCT04003662
Title: Vital Sign Comparison Between Lifelight and Standard of Care - Development
Acronym: VISION-D
Status: Completed | Type: Observational
Sponsor: Xim Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PHT/2018/25 IRAS ID 242581
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Vital Signs
MeSH Terms: interventions — Vital Signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- inpatients: Vital signs measurement - standard of care and prototype
  Interventions: Device: Vital Signs Measurement
- outpatients: Vital signs measurement - standard of care and prototype
  Interventions: Device: Vital Signs Measurement
- Healthy controls: Vital signs measurement - standard of care and prototype
  Interventions: Device: Vital Signs Measurement

INTERVENTIONS:
Device: Vital Signs Measurement — Vital signs are measured twice with standard of care equipment while recording digital video data at the same time.

SUMMARY:
Patients and volunteers both with and without medical problems will be recruited; vital sign measurements are taken twice with normal equipment and while recording video data at the same time. The data collected will allow the Artificial Intelligence to develop the LifeLight algorithm to to improve measurement accuracy of its video data based vital signs monitor.

DETAILED DESCRIPTION:
Vital signs such as heart rate, blood pressure, breathing rate and oxygen levels currently need several pieces of equipment and trained staff in order to be measured properly. The LifeLight app measures the same vital signs using a camera in a phone, tablet, laptop or smart TV. By using very small changes in the colour of your skin, LifeLight's AI system can calculate these values without any extra equipment or training, and without contact.

The aim of this research study is to improve the accuracy of the LifeLight system with a view to a subsequent Validation study to prove the level of accuracy. The investigators will recruit patients, staff and visitors, both with and without medical problems, and take vital sign measurements twice with normal equipment and while recording video data at the same time. This will allow the AI which develops the LifeLight algorithm to make it more accurate, prior to a subsequent study which will validate the results.

ELIGIBILITY:
Inclusion Criteria:

* I1. Sufficiently conversant in the English language to satisfy I3.
* I2. Able and willing to comply with all study requirements.
* I3. Able and willing to provide written informed consent to participate (including by parent or legal guardian if under 16 years old).

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion/exclusion criteria is limited to the proposed intended use of the device, therefore only individuals, of any sex, over the age of 3 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Readings | Single Visit; up to one day
  Comparison of digital video data to standard of care measurement
Oxygen Saturation Readings | Single Visit; up to one day
  Comparison of digital video data to standard of care measurement
Heart Rate (pulse) Readings | Single Visit; up to one day
  Comparison of digital video data to standard of care measurement
Respiratory Rate | Single Visit; up to one day
  Comparison of digital video data to standard of care measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, England, United Kingdom